CLINICAL TRIAL: NCT04387474
Title: China National Clinical Research Center for Neurological Diseases
Brief Title: The Effectiveness of Rehabilitation Training Based on Brain-computer Interface Technology to Improve the Upper Limb Motor Function of Ischemic Stroke.
Acronym: REBUILT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-089-02
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hemiplegia Following Ischemic Stroke
Keywords: Brain-computer interface; Electric stimulation therapy; Stroke rehabilitation
MeSH Terms: interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): brain-computer interface rehabilitation training and traditional rehabilitation training.
  Interventions: Device: Brain-computer interface; Other: Traditional rehabilitation
- Control group (Other): traditional rehabilitation training.
  Interventions: Other: Traditional rehabilitation

INTERVENTIONS:
Device: Brain-computer interface — brain-computer interface rehabilitation training.
  Arms: Experimental group
Other: Traditional rehabilitation — traditional rehabilitation training.

SUMMARY:
To evaluate the effectiveness and safety of rehabilitation training based on brain-computer interface in improving the upper motor function, self-care ability in daily life and quality of life in patients with ischemic stroke. This study adopts centralized uniform random 1:1 grouping, subjects will be randomly assigned to the experimental group and the control group. Randomization schemes are generated by statistical professionals using SAS software.

DETAILED DESCRIPTION:
Brain computer interface(BCI) is a noninvasive nervous system intervention. As a new method, it is applied in rehabilitation by stimulating peripheral nerve, such as motor, vibration, sensory, in combination with other stimulations, such as transcranial magnetic stimulation, transcranial electrical stimulation, etc.

In traditional rehabilitation therapy, hand-holding training is completed by physical therapist. Rehabilitation robot is also used for auxiliary training. BCI therapy will stimulate patients to take part in rehabilitation training more actively and obtain better effects on the rehabilitation of stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (18 years<male or female≤80 years )
2. Ischemic stroke diagnosed by MRI within 1 month before randomization
3. Unilateral upper limb dysfunction with NIHSS score 1-3 at the time of randomization
4. Informed consent signed

Exclusion Criteria:

1. Unable to understand or cooperate because of severe aphasia or cognitive impairment (CDR >0.5) or mental illness
2. A history of epilepsy
3. Sensory disorders or hallucinations
4. Internal carotid artery dissection or thrombolysis
5. Apraxia
6. Agnosia
7. Other diseases that may interfere with motor function
8. Severe cardiopulmonary disease, severe illness, and unstable vital signs
9. Severe balance dysfunction
10. Participating in other clinical trial
11. During pregnancy and lactation
12. The Numerical Rating Scale (NRS) scores of upper extremities>4.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
The improvement of upper limb motor function at 1 month after randomization. | 1 month after randomization compared with traditional rehabilitation strategy.
  Tested by Fugl-Meyer Assessment (FMA) scale.

SECONDARY OUTCOMES:
The improvement of upper limb motor function at 3 month after randomization. | 3 months after randomization compared with traditional rehabilitation strategy .
  Tested by Fugl-Meyer Assessment (FMA) scale.
The improvement of upper limb motor function at 1, 3 month after randomization. | 1, 3 months after randomization compared with traditional rehabilitation strategy.
  Tested by Action Research Arm Test (ARAT), The Wolf Motor Function Test (WMFT).
The improvement in muscle tone at 1, 3 month after randomization. | 1, 3 months after randomization compared with traditional rehabilitation strategy.
  Tested by the Modified Ashworth scale (MAS).
The improvement of patients' ability to take care of themselves in daily life | 1, 3 months after randomization compared with traditional rehabilitation strategy.
  Tested by Instrumental Activity of Daily living (IDAL).

OTHER OUTCOMES:
The changes of brain network properties. | 1 month and 3 months after randomization.
  Evaluated by fMRI before and after rehabilitaion.

CONTACTS AND LOCATIONS:
Locations (1):
- China National Clinical Research Center for Neurological Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
All data described in the outcomes section are available on request to the corresponding author. The protocol and SAP was uploaded in the supplemental materials with the paper

REFERENCES:
- [Derived] Wang A, Tian X, Jiang D, Yang C, Xu Q, Zhang Y, Zhao S, Zhang X, Jing J, Wei N, Wu Y, Lv W, Yang B, Zang D, Wang Y, Zhang Y, Wang Y, Meng X. Rehabilitation with brain-computer interface and upper limb motor function in ischemic stroke: A randomized controlled trial. Med. 2024 Jun 14;5(6):559-569.e4. doi: 10.1016/j.medj.2024.02.014. Epub 2024 Apr 19. PMID 38642555